CLINICAL TRIAL: NCT01396980
Title: Sublingual Microcirculatory Flow Measurements During Haemodialysis in Relation to Blood Volume Change
Brief Title: Microcirculation During Haemodialysis
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, Dr, Frisius Medisch Centrum
Other Study IDs: TPO 776
Record Dates: First submitted 2011-05-31; First posted 2011-07-19 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Complication of Hemodialysis
Keywords: hemodialysis; intensive care; microcirculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dialysis patients: dialysis patients, stabil, dialysis dependancy for more than 3 months, with adequate access

SUMMARY:
* SDF is validated by measuring changes in microcirculation in sepsis patients with MOF (Boerma studies).
* SDF is validated by measuring changes in microcirculation in stable chronic hemodialysis patients (NDT 2009 Bemelmans).
* Ultrafiltration in stable chronic hemodialysis leads to a decrease in sublingual microcirculatory flow (NDT 2009 Bemelmans).
* Trendelenburg position improves the sublingual microcirculatory flow at the end of hemodialysis treatment (NDT 2009 Bemelmans).
* Hemodialysis with ultrafiltration leads to a significant reduction of myocardial perfusion and cardiac output (NDT 2009 Dasselaar)
* Cardiac output measurement during dialysis is not practical.
* BVM is a validated method for hypotension due to ultrafiltration to prevent the amount of ultrafiltration online change based on the measured haemoconcentration (ref Dasselaar et al NDT 2005).
* BCM is a validated measurement to the dry weight in hemodialysis patients measured by a bioimpedance technique (NDT Passauer et al 2009).

DETAILED DESCRIPTION:
The search for an optimal method of ultrafiltration with minimal hypoperfusion of vital organs.

* Stabile hemodialysis patients with dialysis dependancy for more than 3 months, with adequate access
* Study duration 3 weeks
* Number of hemodialysis treatment for purposes of study: 3
* Timing hemodialysis treatments for Study session Monday or Tuesday after the weekend (randomized design in the sessions)

  * session a: 5 hours total duration: 4 hours HD without UF followed by 1 hour GUF
  * Session b: 4 hours total duration: 4 hours HD with UF
  * session c: 4 hours total duration: 4 hours HD with UF and BVM
* UF is determined by actual target weight.
* Measurements during sessions:

  * In each session in advance: blood pressure, pulse, weight, BCM, laboratory tests (Hb, Hct, Na, K, urea, creatinine, calcium, albumin, phosphate, nt-proBNP, troponin T, CRP)
  * During each session at t = 0, t = 1 hour, t =2 hours and t = 4 hours: SDF, blood pressure, pulse, UF at that time, UF rate at that time
  * End each session: blood pressure, pulse, weight, BCM, laboratory tests (Hb, Hct, Na, K, urea, creatinine, calcium, albumin, phosphate, nt-proBNP, troponin T, CRP)

ELIGIBILITY:
Inclusion Criteria:

* dialysis patient
* age > 18
* informed consent

Exclusion Criteria:

* no adequate access
* instable hemodynamics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable hemodialysis patients with dialysis dependancy for more than 3 months, with adequate access
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Difference between sublingual microvascular flow index between 2 types of ultrafiltration | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, MD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands

REFERENCES:
- [Derived] Veenstra G, Pranskunas A, Skarupskiene I, Pilvinis V, Hemmelder MH, Ince C, Boerma EC. Ultrafiltration rate is an important determinant of microcirculatory alterations during chronic renal replacement therapy. BMC Nephrol. 2017 Feb 20;18(1):71. doi: 10.1186/s12882-017-0483-z. PMID 28219329